CLINICAL TRIAL: NCT00684931
Title: Alterations of Fronto-Cerebello-Frontal Loops in Attention Deficit Hyperactivity Disorder (ADHD) : A Study Using Magnetic Resonance Imaging (MRI)
Brief Title: Cerebellar Loops and Attention Deficit Hyperactivity Disorder (ADHD)
Acronym: TDA/H
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in the organisation
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Jean-Pierre LEROY / Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2007/21
Record Dates: First submitted 2008-05-22; First posted 2008-05-28 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention; Deficit; Disorder; Hyperactivity; cerebellum; alteration; fronto-cerebello-frontal loops
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Disease; Spasm | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): patients with Attention Deficit Disorder with or without Hyperactivity
  Interventions: Other: Imaging
- 2 (Sham Comparator): healthy volunteer without Attention Deficit Hyperactivity Disorder
  Interventions: Other: Imaging

INTERVENTIONS:
Other: Imaging — neuropsychological evaluation and Imaging with magnetic resonance (MRI)

SUMMARY:
The aim of this study is to investigate the integrity of connectivity between the neocortex and the cerebellum in the Attention Deficit Hyperactivity Disorder (ADHD). Fibers integrity will be measured using magnetic Resonance Imaging Techniques.

DETAILED DESCRIPTION:
ADHD is a neurodevelopmental trouble characterized by attentional deficits, impulsivity and motor hyperactivity. Morphological neuroimaging studies in ADHD children have revealed cerebellar abnormalities, however data in adults regarding cerebellum alterations are scarce. In this study we will analyse the conectivity of the cerebellum of adults ADHD patients. We will use diffusion tensor imaging (DTI) technique, and morphological data will be compared with the neuropsychological status.

ELIGIBILITY:
Inclusion Criteria:

Patient with ADHD :

* Diagnosis of ADHD
* 18 - 35 years old

Healthy volunteer :

* 18 - 35 years old
* no ADHD diagnosed

Exclusion Criteria:

* Associated neurological or psychiatric pathologies
* Pregnant woman
* MRI counter indication

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2008-02; Primary Completion 2008-02 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Fractional anisotropy coefficient if fronto-cerebello-frontal loops. | visite 1

CONTACTS AND LOCATIONS:
Overall Officials: Manuel BOUVARD, MD, Principal Investigator — Charles Perrens Hospital
Locations (2):
- France (2):
  - Charles Perrens Hospital, Bordeaux
  - University Hospital Bordeaux, Bordeaux